CLINICAL TRIAL: NCT00780845
Title: AKIN (Acute Kidney Injury Network): Acute Kidney Injury After On-Pump Coronary Artery Bypass Graft Surgery
Brief Title: AKIN Criteria: Acute Kidney Injury After On-Pump Coronary Artery Bypass Graft (CABG)
Status: Completed | Type: Observational
Sponsor: Hospital de Base (Other)
Responsible Party: Mauricio N Machado, São José do Rio Preto Medical School
Other Study IDs: CAAE-3438.0.000.140-08
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-10

CONDITIONS: Kidney Failure
Keywords: Acute Kidney failure; Clinical outcomes; On-pump; Coronary artery bypass grafting; Morbidity; Mortality
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI (-): Patients without acute kidney injury after on-pump CABG
- AKI (+): Patients with acute kidney injury after on-pump CABG

SUMMARY:
The purpose of this study is evaluate clinical outcomes and 30-day mortality after on-pump CABG.

DETAILED DESCRIPTION:
Eight hundred and seventeen patients was enrolled in this series and divided into to groups: Group AKI (-) - patients without acute kidney injury after on-pump CABG. Group AKI (+) - patients with acute kidney injury after on-pump CABG. AKI was defined as an absolute increase in serum creatinine (SCr) of more than or equal to 0.3 mg/dl (≥ 26.4 μmol/l) or a percentage increase in SCr of more than or equal to 50% (1.5-fold from baseline). The change in SCr concentration was defined as the difference between immediate postoperative concentration and the highest concentration during the stay in ICU. Clinical Outcomes and 30-day mortality was evaluate in this patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent on-pump coronary artery bypass grafting
* Patients with at least two serum creatinine values within 48 hours.

Exclusion Criteria:

* Patients with end-stage kidney disease requiring renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups AKI (-) and AKI (+) selected consecutively after admission in cardiac surgery postoperative care unit
Sampling Method: Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that patients with acute kidney injury after on-pump CABG have higher 30-day mortality | 30 days

SECONDARY OUTCOMES:
To compare clinical outcomes in patients with and without acute kidney injury after on-pump CABG | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lilia N Maia, PhD, Study Director — São José do Rio Preto Medical School

REFERENCES:
- [Derived] Machado MN, Miranda RC, Takakura IT, Palmegiani E, Santos CA, Oliveira MA, Mouco OM, Hernandes ME, Lemos MA, Maia LN. Acute kidney injury after on-pump coronary artery bypass graft surgery. Arq Bras Cardiol. 2009 Sep;93(3):247-52. doi: 10.1590/s0066-782x2009000900008. English, Portuguese, Spanish. PMID 19851652